CLINICAL TRIAL: NCT07090226
Title: Assessing Spatial Frequency Domain Imaging as an Objective Quantification of Longitudinal Skin Changes in Scleroderma
Brief Title: Diffuse Cutaneous Scleroderma (DSSc) SFDI Study
Acronym: SFDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-46158; R01AR085317-01 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Systemic Scleroderma; Diffuse Cutaneous Scleroderma
Keywords: Spatial frequency domain imaging (SFDI); modified Rodnan skin score (mRSS); Skin biopsy; Skin fibrosis; Scleroderma skin patient reported outcome (SSPRO); Durometry; Ultrasound; Diffuse cutaneous scleroderma (dcSSc)
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: There will be 60 patients with scleroderma and 5 control participants without scleroderma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scleroderma Participants (Experimental): Participants in this arm will be asked to complete the Fitzpatrick skin type questionnaire to quantify skin tone and will have measurements taken with a colorimeter on the right and left forearms, hands, and fingers to quantify skin tone. At each study visit, a physician will measure the mRSS and take SFDI measurements. Ultrasound and durometry will then be done. Optional skin biopsies will be collected from the forearm at baseline and 12 months.
  Interventions: Other: Spatial-frequency domain imaging (SFDI)
- Control (Active Comparator): Participants in this arm will be asked to complete SFDI and colorimeter measurements.
  Interventions: Other: Spatial-frequency domain imaging (SFDI)

INTERVENTIONS:
Other: Spatial-frequency domain imaging (SFDI) — SFDI is a method using near-infrared (NIR) light to generate wide field images (>10 x 10 cm) of tissue optical properties (absorption and scattering coefficients) at sub-surface depths of 1-10 mm. With SFDI the tissue surface (skin) is illuminated by a rapid sequence of sinusoidal light patterns of varying spatial frequency and at different optical wavelengths. Collected camera images are then processed to yield maps of sub-surface optical properties.

SUMMARY:
Scleroderma (SSc) is an autoimmune disease characterized by fibrosis (or collagen deposition) of the skin and internal organs. The extent of skin fibrosis is an important predictor of internal organ complications and increased mortality. Currently a very imprecise, subjective method that varies amongst different doctors for the same patient is used to quantify skin fibrosis in patients, by "pinching" their skin and assessing how thick it is; this is the method used to determine the modified Rodnan skin score (mRSS).

A previous plot study was conducted by the investigators to determine if spatial frequency domain imaging (SFDI), a method of light scattering, could be used to measure the collagen content in the skin of SSc patients. This non-painful, noninvasive method takes very little time and the investigators hypothesized that it would be more accurate than the "pinching" method. For that pilot study, patients with various stages of the disease were selected, and SFDI was used to image 6 areas. A forearm skin biopsy was taken for subsequent histopathology analyses of collagen content. The clinical mRSS was assessed at the time of SFDI measurement. Optical property imaging data was analyzed and statistically correlated and analyzed with immunohistochemistry (a method of identifying proteins) of the skin. Preliminary results demonstrated a strong correlation between mRSS and SFDI. Some of the imaging parameters of the SFDI were modified based on the initial results. Initial results demonstrated that the device can detect increases in skin thickness observed in SSc skin.

DETAILED DESCRIPTION:
* The primary objective of this study is to validate spatial-frequency domain imaging (SFDI) and related optical techniques as robust, sensitive, and objective methods for quantifying skin involvement in systemic sclerosis. The study aims to use SFDI/SLIM to examine longitudinal skin changes in early diffuse cutaneous SSc patients and the correlation with change in modified Rodnan Skin Score (mRSS).
* Secondary objectives include assessing correlations between SFDI measurements of skin in SSc subjects and other clinical outcomes such as durometry, ultrasound, histopathological changes in the skin, or scleroderma patient reported outcomes (PROs).

In the current study longitudinal measurements in SSc patients will be taken to examine: the sensitivity and accuracy of SFDI to detect changes in skin thickness over time in response to therapy or from disease progression, the correlation between SFDI measurements and mRSS, and the expression of proteins including PDGFRβ in skin biopsy tissue.

In this study SFDI and other clinical outcome assessments of skin thickness and fibrosis in scleroderma patients including skin biopsy histology, scleroderma skin patient reported outcome (SSPRO), ultrasound, and durometry (durometer measures skin hardness) will be compared. SFDI information will also be compared with capillaroscopy (that allows for non-invasive imaging of the nailfold capillaries) if available from the electronic medical record. If SFDI correlates well with other clinical outcome assessments, it may be used as a rapid, non-invasive tool for monitoring disease activity in scleroderma patients.

ELIGIBILITY:
Inclusion Criteria:

* Scleroderma (SSc) participants must have been diagnosed with SSc as defined by the American College of Rheumatology within the past 2-5 years AND fulfill criteria for diffuse cutaneous SSc according to LeRoy classification
* Healthy controls must be free of SSc or other autoimmune disease and have no known skin pathology

Exclusion Criteria:

* Diagnosis of skin malignancy within the previous 2 years, excluding adequately treated squamous cell skin cancer, basal cell carcinoma, and carcinoma in situ.
* Presence of wounds or skin rashes at the site of Spatial frequency domain imaging (SFDI) measurement or skin biopsy
* Presence of other co-morbid illnesses with an estimated median life expectancy < 5 years.

Exclusion criteria for providing a skin biopsy sample during the study but are not exclusions for enrollment in the study.

* Subject has known allergy to lidocaine or has had a reaction to local anesthetics in the past will not provide skin biopsy samples at any time during the study.
* Subjects who, in the opinion of the investigator, are high-risk for small tissue calcification, or other conditions that may affect wound healing will not provide skin biopsy samples at any time during the study.
* Subjects who are pregnant or lactating are excluded from providing a skin biopsy sample only while they are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Spatial-frequency domain imaging (SFDI) measurements of skin thickness | Baseline, 3 months, 6 months.12 months
  SFDI measurements will be obtained on the right and left fingers, hands, and upper arms and forearms. Total SFDI score is defined as the sum of the individual SFDI measurements.
Modified Rodnan skin score (mRSS) measurements of skin thickness | Baseline, 3 months, 6 months.12 months
  One of two methods will be used to assess the mRSS: 1) gently pinch the skin using the index finger and thumb, or 2) press the skin between two thumbs to form a fold of skin. to score the 17 body areas on a scale. of 0-3 (0 is normal, 1 is mild thickness, 2 is moderate thickness, and 3 is severe thickness). The range of possible scores is 0 to 51 and a higher total mRSS score generally indicates more severe skin involvement and a worse prognosis in SSc.

SECONDARY OUTCOMES:
Ultrasound measurements of the forearms | Baseline, 3 months, 6 months.12 months
  A high frequency ultrasound scanner (GE Logiq e) with a 20 MHz transducer will be used to assess dermal thickness. Dermal thickness will be defined as the distance between the dermal-epidermal junction and the dermal-subcutaneous tissue interphase. Measurements will be taken at both the right and left border and the mean of these will be recorded as the dermal thickness score.
Ultrasound measurements of the hands | Baseline, 3 months, 6 months.12 months
  A high frequency ultrasound scanner (GE Logiq e) with a 20 MHz transducer will be used to assess dermal thickness. Dermal thickness will be defined as the distance between the dermal-epidermal junction and the dermal-subcutaneous tissue interphase. Measurements will be taken at both the right and left border and the mean of these will be recorded as the dermal thickness score.
Ultrasound measurements of the fingers | Baseline, 3 months, 6 months.12 months
  A high frequency ultrasound scanner (GE Logiq e) with a 20 MHz transducer will be used to assess dermal thickness. Dermal thickness will be defined as the distance between the dermal-epidermal junction and the dermal-subcutaneous tissue interphase. Measurements will be taken at both the right and left border and the mean of these will be recorded as the dermal thickness score.
Durometry measurements of the forearm | Baseline, 3 months, 6 months.12 months
  Skin hardness will be measured using a hand-held digital durometer (Rex Gauge type OO; Rex Gauge, Buffalo Grove, IL). Three consecutive measurements will be taken at each forearm (center of dorsal aspect, midway between the radial head/styloid and lateral epicondyle). The mean of the 3 measurements at each site will be used.
Durometry measurements of the hands | Baseline, 3 months, 6 months.12 months
  Skin hardness will be measured using a hand-held digital durometer (Rex Gauge type OO; Rex Gauge, Buffalo Grove, IL). Three consecutive measurements will be taken at each hand. The mean of the measurements at each site will be used.
Collagen content of the forearm | Baseline, 12 months
  Trichrome staining of a skin biopsy will be done to assess collagen content.
Scleroderma patient reported outcomes (SSPRO) scores | Baseline, 3 months, 6 months.12 months
  The SSPRO is a self-administered 18 item questionnaire to assess the effects of skin changes on physical, emotional and social well-being of SSc patients. Each question is rated on a scale from 0 (not much) to 6 (very much) with the maximum score being 108. Higher scores are associated with more adverse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Bujor, MD, PhD, Principal Investigator — BU Chobanian & Advesian School of Medicine
Locations (1):
- Shapiro Outpatient Rheumatology Clinic at Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No